CLINICAL TRIAL: NCT02665702
Title: Endostar Combined With NVB and DDP Second-line Treatment of Advanced Esophageal Squamous Cell Carcinomas of the Prospective, Single Arm Phase II Clinical Study
Brief Title: Endostar Combined With NVB and DDP Second-line Treatment of Advanced Esophageal Squamous Cell Carcinomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-SH-001
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Vinorelbine; Cisplatin; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar Combined With NVB and DDP (Experimental): Endostar15mg/m2 NVB25 mg/m2 DDP75 mg/m2
  Interventions: Drug: NVB; Drug: DDP; Drug: Endostar

INTERVENTIONS:
Drug: NVB — 25mg/m2 ，D1，8
  Other Names: Vinorelbine Injection
Drug: DDP — 75mg/m2 ，D1 or 25mg/m2 D1-3
  Other Names: Cisplatin
Drug: Endostar — 15mg/d，d1-d7 civ
  Other Names: endo

SUMMARY:
The aim of this study is to explore whether endostar combined with NVB and DDP as treatment could improve progression-free surial time (PFS) and to evaluate the safety of the chemotherapy regimens

DETAILED DESCRIPTION:
This study is to explore whether endostar combined with NVB and DDP as treatment could improve progression-free surial time (PFS) and to evaluate the safety of the chemotherapy regimens used as second-line treatment of advanced esophageal squamous cell carcinomas

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary thoracic esophageal squamous cell carcinoma
2. According to the esophageal AJCC2009 7th to determine new stage IV esophageal cancer
3. The subject has PD after first-line chemotherapy or radiation within a year
4. Presence of at least one index lesion measurable by CT scan or MRI according to RECIST 1.1
5. Can eat more than liquid diet; No signs before esophageal perforation
6. 18~75 years
7. PS:0-1
8. Life expectancy of ≥ 3 months
9. ANC ≥ 2×109/L，PLT ≥ 100×109/L，Hb ≥ 90g/L
10. TB ≤ UNL； ALT/AST ≤ 2.5×UNL，AKP ≤ 5×UNL
11. Ccr≤ UNL,Scr≥60 mL/min
12. Normal electrocardiogram (ecg), the body had no unheal wounds
13. Radiotherapy before within the scope of the normal dose and not affect subsequent treatment
14. Prior to biological agents, especially e. coli genetically engineered products without severe allergic reactions
15. Signed written informed consent

Exclusion Criteria:

1. Breast-feeding or pregnant women, no effective contraception if risk of conception exists
2. Chronic diarrhea, enteritis, intestine obstruction which are not under control
3. Esophageal obstruction cannot eat liquid completely, esophagus have deep ulcer perforation or hematemesis; Esophageal cancer common complications such as anastomotic leakage, serious lung complications, etc.
4. A second primary tumor (except skin basal cell carcinoma)
5. The original serious heart disease, including: higher risk of congestive heart failure, unable to control arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension
6. With uncontrol nerve, mental illness or mental disorders, compliance is poor, can't cooperate with accounts and response to treatment; Primary brain tumors or CNS metastases illness did not get a control, has obvious cranial hypertension or nerve mental symptoms
7. With bleeding tendency
8. Has inherited bleeding evidence of physical or blood coagulation disorder
9. With clear chemotherapy drug allergy
10. Other researchers believe that patients should not participate in this testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided